CLINICAL TRIAL: NCT02067585
Title: An Analysis of Lipid and Glucose Metabolism Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008986; Edmonton Civic Employees (Other Grant/Funding Number: Edmonton Civic Employees)
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAGB (Experimental): Standardized Lipid meals will be served to Laparoscopic adjustable gastric banding patients.
  Interventions: Dietary Supplement: Standardized Lipid meals
- LRYGB (Experimental): Standardized Lipid meals will be served to the Laparoscopic Rou-en-Y gastric bypass patients.
  Interventions: Dietary Supplement: Standardized Lipid meals
- Non-surgical (Experimental): Standardized Lipid meals will be served to the non-surgical obese patients
  Interventions: Dietary Supplement: Standardized Lipid meals

INTERVENTIONS:
Dietary Supplement: Standardized Lipid meals — Standardized Lipid meals: 240 ml of Hormel Great Shake Plus liquid nutritional supplement, 203 Kcal/100mL; 49% calories from fat, mostly unsaturated fatty acids of soy origin; 38% calories from carbohydrates, 13% calories from proteins.

SUMMARY:
Bariatric surgery induce remarkable weight loss and improvement or resolution of type 2 diabetes. Obesity is the primary risk factor for type 2 diabetes, and 90% of all type 2 diabetics are obese. Type 2 diabetes resolves post-operatively in 84-98% after bypass and 48-68% after restrictive procedures.

Obesity leads to elevated plasma free fatty acids and subsequently to excessive accumulation of triglyceride in peripheral tissues, which is an independent risk factor for insulin resistance and type 2 diabetes. Bariatric surgery is associated with dramatic decrease in plasma free fatty acids and other lipids.

This study will clarify the relationship of changes in fatty acid and other lipid metabolism to improved insulin sensitivity after different bariatric procedures ('restrictive' - laparoscopic adjustable gastric band and 'hybrid' - laparoscopic roux-en-y gastric bypass) and compare them with non-surgical obese patients. This will allow the investigators to refine indications for these procedures especially in patients with type 2 diabetes.

The investigators will analyze whether surgical bypass of the upper small bowel plays a critical role in the resolution of type 2 diabetes and improvement in lipid metabolism. The investigators will achieve this by comparing gastric banding and gastric bypass in a collaborative research study involving obesity surgeons, physicians and lipid researchers.

DETAILED DESCRIPTION:
Background: Bariatric surgery is the only evidence-based approach to efficacious and sustainable weight loss. It is estimated that about one third of patients undergoing bariatric surgery have type 2 diabetes, with a high rate of resolution of diabetes post-operatively: 84-98% after gastric bypass and 48-68% after purely restrictive procedures(1, 2). Other cardiovascular risk factors such as lipid profile and inflammatory markers also, significantly improve. 25% of the population of Alberta are obese and 2,7% are morbidly obese, one third of them are with type 2 diabetes. Bariatric surgery in these patients will translate into a cure for type II diabetes, dramatic improvements in quality of life, improved longevity and lower health care costs for the system.

Morbid obesity leads to elevated plasma free fatty acids (FFA) and subsequently to excessive accumulation of triglyceride in peripheral tissues. Excessive triglyceride accretion is an independent risk factor for insulin resistance, type II diabetes and cardiovascular complications. Bariatric surgery is associated with dramatic improvements in these comorbid diseases(2). Purely restrictive procedures (laparoscopic adjustable gastric band - LAGB) may differ from hybrid procedures (laparoscopic roux-en-y gastric bypass - LRYGB) in their effect on diabetes and cardiovascular disease. The LAGB is a less complex surgical procedure that can be done on a day surgery basis and has an extremely low peri-operative mortality rate. The LRYGB is much more complex and has a low but important rate of anastomotic leak and mortality.

LAGB and LRYGB vary in their average percent excess weight loss (%EWL)(2). This may contribute to a disparity in their impact on comorbid disease. However, improvements in insulin sensitivity and glucose homeostasis occur early after LRYGB, preceding significant weight loss(3). Postoperative changes in the absorption and metabolism of lipids induced by a malabsorptive procedure may be responsible for these beneficial changes. The relationship of improved insulin sensitivity to changes in lipid metabolism need to be clarified in order to understand the varying impact of LAGB and LRYGB on comorbid disease associated with obesity. The initial decreased caloric intake following Bariatric surgery can improve the response of adipose tissue manifested by favorable changes in adipocytokines. The postoperative rise in adiponectin (4, 7) (an anti-inflammatory mediator) was observed. These changes correlate with weight loss and improvement in insulin resistance.

In obese insulin-resistant subjects, insulin cannot attenuate hydrolysis of stored triglyceride in adipose tissue and consequently this leads to excessive free fatty acids release into circulation and increased delivery of fatty acids to the muscle, liver and pancreas. Excessive uptake of fatty acids into these tissues exacerbates hepatic and muscle insulin resistance and impairs insulin secretion from pancreatic beta cells. Bariatric surgery improves insulin sensitivity which leads to inhibition of hydrolysis of adipose triglycerides and decreased release of free FFA into the circulation. Recently it was shown that not only increased baseline FFA but also altered clearance of FFA normalize after LRYGB (8). Also, postoperative reduction in fat intake and absorption leads to decreased level of FFA in blood. After malabsorptive, weight-reducing procedures the beta cell glucose and fatty acid sensitivity was doubled early in diabetic patients, leading to a decrease in insulin secretion (9).

Beside its contribution to insulin resistance, severe obesity is also associated with an elevated inflammatory state. In obese with type 2 diabetes and metabolic syndrome, the highly sensitive C-reactive protein (CRP) serum concentration, an inflammatory marker, is increased and correlates with the severity of glucose intolerance and with the severity of inflammation (10). Following bariatric surgery, C-reactive protein (CRP) decreases. It has been shown that gastric bypass reduces biochemical cardiac risk factors, particularly, CRP by 80% in addition to triglycerides, total cholesterol, LDL, and lipoprotein A (7, 11).

These changes in lipid and glucose metabolism are seen after restrictive and hybrid procedures to a varying extent. Given the different mechanism of action, technical complexity and safety profiles of LAGB and LRYGB, it is crucial to clarify their impact on co-morbid disease.

Hypothesis:

1. Postprandial reduction in serum levels of free fatty acids and lipids following LRYGB (a malabsorptive procedure) are greater than following LAGB (a purely restrictive procedure).
2. Reduced serum levels of free fatty acids and lipids following LRYGB lead to improvements in insulin resistance.

Rationale: Clinical evidence suggests that purely restrictive procedures (LAGB) affect lipid absorption and metabolism differently when compared to hybrid restrictive/malabsorptive procedures (LRYGB). This may be due to the malabsorptive component of LRYGB where ingested food bypasses the duodenum and upper jejunum, both important for lipid digestion and absorption.

Design: A cross-sectional study to characterize lipid absorption and metabolism following bariatric surgical procedures based out of the Weight Wise Clinic at the Royal Alexandra Hospital, Edmonton. Venous blood will be collected after overnight fast, before and after standardized lipid meal, and analyzed for appropriate biochemical indices. The study cohorts will comprise patients after LAGB, LRYGB, in the period of weight stabilization, 12+ months following bariatric surgery. Controls will comprise preoperative patients managed without pharmacologic intervention for their obesity.

Methods: Recruitment and physical examination will be conducted at the Weight Wise Clinic. Studies will begin at the Clinical Investigation Unit, University of Alberta Hospital, at 7 AM after a consumed the night before study meal and then 12-h-overnight fast. Liquid meal will consist of 240 ml of Hormel Great Shake Plus liquid nutritional supplement, 203 Kcal/100mL; 49% calories from fat, mostly unsaturated fatty acids of soy origin; 38% calories from carbohydrates, 13% calories from proteins. Weight measurement will be performed by a nurse. Fasting baseline blood will be drawn and the subjects will consume a second portion of the study meal. The test meal will be drunk with a straw within 15 minutes. Blood withdrawal will be carried out at 10, 20, 30, 90 min, 4 and 6 hrs after the start of ingestion of the standardized meal. Subjects will be allowed to walk or sit, but not to exercise during the test. Drinking of water without sugar will be permitted. Blood will be collected through a venous in-dwelling catheter placed in a cubital vein.

Laboratory analyses: The plasma total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglycerides, nonesterified fatty acid concentration and the degree of unsaturation, ApoB-48 (intestinally-derived lipoprotein) and apoB-100 (liver-derived lipoprotein), insulin, glucose, CPR, adiponectin, HbA1c, albumin, AST, ALT, ketone bodies will be measured.

Primary outcome: postprandial changes in serum free fatty acids, lipids (cholesterols total, LDL and HDL, triglycerides) and apoB in patients after bariatric surgery and their relationship with insulin sensitivity (glucose, insulin, HOMA index).

The investigators expect that greater reduction in postprandial serum free fatty acids and lipids (cholesterol, triglyceride) after LRYGB will be associated with greater decrease in insulin resistance (HOMA index is expected to decrease), as compared with LAGB. Insulin, plasma glucose and ketone bodies are expected to decrease.

Secondary outcomes: Changes in HbA1c, AST, ALT, albumin, CRP, adiponectin levels will be compared with the changes in fatty acids, lipids and insulin resistance.

The investigators expect that reduced serum free fatty acid level will be associated with decrease in marker of inflammation (CRP), HbA1c, AST, ALT, and increase in anti-inflammatory mediator (adiponectin) after both procedures, but more pronounced after LRYGB.

Sample Size Calculation: Sample size was calculated based on review of literature showing decrease in post-bariatric procedure free fatty acids. A power analysis was performed with a beta of 0.20 and an alpha of 0.05. Assuming that a 30% difference in the level of FFA exists between morbidly obese operated and not operated patients, 16 subjects will need in each arm, total 48 for LAGB, LRYGB and control groups. Thus the study would provide an 80% chance that a difference would be detected if one exists.

Data analysis: Multivariate Analysis for testing statistical significance of improved serum free fatty acid, ApoB and lipid levels and their correlation with insulin sensitivity (glucose, insulin) among multiple groups of data will be performed by a statistician.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients
* age 18-65
* with or without type 2 diabetes
* 12 or more months following LRYGB or LAGB, or patients waiting for mentioned procedures
* able to provide written informed consent.

Exclusion Criteria:

* chronic liver disease
* maladaptive eating behavior
* current pharmacological treatment for obesity
* for patients following LAGB - ongoing band volume adjustments
* hypothyroidism
* treatment with insulin
* revision of a previous bariatric procedure
* major postoperative complication
* allergy to soy or any component of the study meal
* renal failure (glomerular filtration <60mL/min)
* alcoholism
* acute illness
* pregnancy or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Birch, MD, Principal Investigator — CAMIS, University of Alberta
Locations (1):
- CAMIS, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: no-operated
Period: Overall Study
Arm/Group | LAGB | LRYGB | Control
Started | 16 | 16 | 16
Completed | 16 | 16 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Standardized Lipid meals will be served to the no-operated patients.
  Standardized Lipid meals: Standardized Lipid meals: 240 ml of Hormel Great Shake Plus liquid nutritional supplement, 203 Kcal/100mL; 49% calories from fat, mostly unsaturated fatty acids of soy origin; 38% calories from carbohydrates, 13% calories from proteins.
- Total: Total of all reporting groups
Arm/Group | LAGB | LRYGB | Control | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9) | 48 (10) | 46 (9) | 46 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 15 | 42
  Male | 4 | 1 | 1 | 6
weight current [Mean (Standard Deviation); unit: kg] | 108.7 (26.4) | 108.5 (21.1) | 115.8 (17.1) | 111.0 (21.7)
waist circumference [Mean (Standard Deviation); unit: cm] | 118 (16) | 121 (16) | 122 (8) | 121 (14)
Type 2 diabetes [Count of Participants; unit: Participants] | 2 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Triglycerides Post-prandial
Time Frame: 0 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 95 (64) | 71 (53) | 134 (92)

2. Primary Outcome: Triglycerides
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 93 (64) | 85 (71) | 115 (79)

3. Primary Outcome: Triglyceride
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 123 (75) | 87 (61) | 174 (101)

4. Primary Outcome: Triglyceride
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 124 (93) | 72 (63) | 182 (150)

5. Primary Outcome: Triglyceride
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 103 (67) | 59 (51) | 123 (87)

6. Secondary Outcome: Blood Glucose
Time Frame: 0 minute
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 4.8 (0.4) | 4.7 (0.4) | 5.5 (0.9)

7. Secondary Outcome: Glucose
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 5.3 (0.7) | 7.4 (1.6) | 6.2 (1.1)

8. Secondary Outcome: Glucose
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 5.3 (0.7) | 3.8 (0.8) | 5.9 (1.9)

9. Secondary Outcome: Glucose
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 4.7 (0.5) | 4.6 (0.4) | 5.1 (0.9)

10. Secondary Outcome: Glucose
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LAGB | LRYGB | Control
Number analyzed (Participants) | 16 | 16 | 16
mmol/L | 4.8 (0.9) | 4.7 (0.3) | 4.9 (0.4)

ADVERSE EVENTS:
Arm/Group | LAGB | LRYGB | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 5/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAGB (N=16) | LRYGB (N=16) | Control (N=16)
Mild nausea (Gastrointestinal disorders) | 0 | 2 | 1
Mild headache (General disorders) | 0 | 1 | 1
Blood Glucose < 3mmol/L (90 mins post-meal) (Endocrine disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No